CLINICAL TRIAL: NCT02716480
Title: Impact of the Use of Health-connected Devices on Recovery of Physical Activity in Obese Patients After Bariatric Surgery.
Brief Title: Health-connected Devices and Physical Activity Recovery in Bariatric Surgery Patients
Acronym: MYGOODTRIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: My Goodlife SAS (Industry)
Collaborators: European Georges Pompidou Hospital (Other); Hospital Ambroise Paré Paris (Other); French Environment and Energy Management Agency (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MY GOODLIFE
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate
Keywords: Nutrition; Physical activity; Bariatric surgery; Obesity; Health technology; Health-connected devices
MeSH Terms: conditions — Obesity, Morbid; Motor Activity; Obesity | interventions — Range of Motion, Articular; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobility Coaching (Experimental): 45 patients undergoing bariatric surgery received a monthly "mobility" coaching session of 20 to 30 min by phone during 6 months.
  Interventions: Behavioral: Mobility coaching
- Diet Coaching (Experimental): 45 patients undergoing bariatric surgery received a monthly "diet" coaching session of 20 to 30 min by phone during 6 months.
  Interventions: Behavioral: Diet coaching

INTERVENTIONS:
Behavioral: Mobility coaching — The intensive follow-up for the patients of "Mobility Coaching " arm will consist on a monthly remote coaching of 20 to 30 minutes led by a "Mobility" coach. The web platform allows self-administration of a questionnaire to establish patient's diagnosis of mobility to enable personalized coaching. The web platform can also track the parameters collected by connected devices (pedometer and connected scale), organize appointments with patients and ensure the traceability of exchanges with patients. A smartphone application tracks different modes of locomotion used.
  Other Names: Mobility
  Arms: Mobility Coaching
Behavioral: Diet coaching — The intensive follow-up for the patients of "Diet Coaching " arm will consist on a monthly remote coaching of 20 to 30 minutes led by dietitian trained in the care of patients undergoing bariatric surgery.
  Other Names: Diet
  Arms: Diet Coaching

SUMMARY:
The goal of clinical trial is to evaluate the impact of use of health-connected devices and of an Internet-based Intensive follow-up on physical activity recovery during the 6-month period after bariatric surgery in obese patients.

DETAILED DESCRIPTION:
90 patients with morbid obesity, having recently benefited from an act of bariatric surgery will be recruited for clinical trial if they meet the inclusion and no inclusion criteria. This is a single-center, open, controlled, randomized, 2 parallel-groups:

* "Mobility Coaching" group
* "Diet Coaching" group

The "Diet Coaching" group will be the "control group" of "Mobility Coaching" group and vice versa.

Patients in both groups will be equipped with a connected-scale and a wristwatch equipped with a pedometer connected. The online tools available to patients will be used to motivate patients to progress and alert the coaches and the medical team in case of difficulties to achieve the objectives.

ELIGIBILITY:
Inclusion Criteria:

* Primo-surgery bariatric surgery a week before their inclusion
* Absence of surgical side events related to the surgical procedure
* Adult female or male
* Weight ≤ 150 kg
* Knowing read and write French routinely,
* Possessing an internet connection at home,
* Possessing and knowing how to use a computer or tablet,
* Owning a smartphone,
* Affiliated with a social security scheme
* Not Trust
* Having signed the informed consent letter

Non-inclusion criteria • Patient with major disabilities causing a definitive loss of mobility

Exclusion Criteria:

• None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06; Primary Completion 2018-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline mean number of steps per day at 6th month | Period from Day 164 to Day 179
  The primary endpoint is the difference between mean number of steps recorded by the pedometer during the last 15 days of the 6th month (Period Day 164 to Day 179) and the mean number of steps per day recorded in the last 15 days of the first month (Period Day 15 to Day 30).
  .

SECONDARY OUTCOMES:
Change from baseline mean daily energy expenditure at 6th month | At 6th month
  Estimated by self-administrated questionnaire (RPAQ)
Change from baseline mean daily energy expenditure at 3rd month | At 3rd month
  Estimated by self-administrated questionnaire (RPAQ)
Change from baseline weight at 6th month | At 6th month
Change from baseline weight at 3rd month | At 3rd month
% of patients having nutritional deficiency in vitamins and / or minerals | At 6th month
  Biological measurements
Change from baseline Quality of life at 6th month | At the 6th month
  Estimated by self-administered quality-of-life questionnaire (EQVOD)
Change from baseline Quality of life at 3rd month | At the 3rd month
  Estimated by self-administered quality-of-life questionnaire (EQVOD)
Change from baseline mean number of steps per day at 3rd month | Period from Day 75 to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Karl AUZOU, Msc, Study Director — My Goodlife SAS
Locations (1):
- Department of Visceral Surgery - European Georges Pompidou Hospital -, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blood Pressure Lowering Treatment Trialists' Collaboration; Ying A, Arima H, Czernichow S, Woodward M, Huxley R, Turnbull F, Perkovic V, Neal B. Effects of blood pressure lowering on cardiovascular risk according to baseline body-mass index: a meta-analysis of randomised trials. Lancet. 2015 Mar 7;385(9971):867-74. doi: 10.1016/S0140-6736(14)61171-5. Epub 2014 Nov 4. PMID 25468168
- [Background] Thereaux J, Corigliano N, Poitou C, Oppert JM, Czernichow S, Bouillot JL. Comparison of results after one year between sleeve gastrectomy and gastric bypass in patients with BMI >/= 50 kg/m(2). Surg Obes Relat Dis. 2015 Jul-Aug;11(4):785-90. doi: 10.1016/j.soard.2014.11.022. Epub 2014 Dec 4. PMID 25771441
- [Result] Czernichow S, Moszkowicz D, Szwarcensztein K, Emery C, Lafuma A, Gourmelen J, Fagnani F. Impact of bariatric surgery on the medical management and costs of obese patients in France: an analysis of a national representative claims database. Obes Surg. 2015 Jun;25(6):986-96. doi: 10.1007/s11695-014-1488-3. PMID 25366293
- [Derived] Lurbe I Puerto K, Bruzzi M, Rives-Lange C, Poghosyan T, Bretault M, Chatellier G, Vilfaillot A, Chevallier JM, Czernichow S, Carette C. MyGood Trip, a Telemedicine Intervention for Physical Activity Recovery After Bariatric Surgery: Randomized Controlled Trial. JMIR Form Res. 2023 Mar 28;7:e26077. doi: 10.2196/26077. PMID 36976624